CLINICAL TRIAL: NCT05777122
Title: Assessing the Effective Method of Pain Reduction After the Placement of Conventional Separators
Brief Title: Pain Reduction After Separators Placement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sadaf Bashir (Other)
Responsible Party: Sponsor-Investigator, Sadaf Bashir, assessing the effective method of pain reduction after the placement of conventional separators, Karachi Medical and Dental College
Organization: Karachi Medical and Dental College (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMDC/COD/ESRC/0047/2021
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Orthodontic Pain
Keywords: pain reduction ,separator, chewing gum, lignocaine gel, VAS
MeSH Terms: interventions — Forkhead Box Protein M1

STUDY DESIGN:
Intervention Model Description: In our study all the participant were asked to fill the questionnaire.In the topical gel group the patients were directed to apply the gel on the buccal free gingival margin of their first molar at one side when the separators are placed and reapply the gel every 8 hours . T'hey were then requested to mark their level of pain at 2 and 8 hours and at 10 pm of the 2nd,3rd,5th and 7th day after the gel is being applied and mark it on the VAS form.
  The patients in the chewing gum group were advised to chew sugar free gum for 5 minutes immediately after separators were placed and at 8 hours interval. The patients were also advised and motivated not to take any additional analgesics.For measuring the perception of pain the most reliable method the Visual Analog Scale (VAS).will be used
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): lignocaine gel every 8 hours
  Interventions: Drug: lignocaine gel
- group B (Experimental): chewing gum every 8 hours 5-10 mins chew
  Interventions: Other: sugar free chewing gum

INTERVENTIONS:
Drug: lignocaine gel — pharmacological ,topical anesthetic gel
  Other Names: somogel
  Arms: group A
Other: sugar free chewing gum — non pharmacological
  Other Names: trident
  Arms: group B

SUMMARY:
Rationale of study:

Separators placement is the primary step in orthodontic treatment and it is almost always accompanied by pain and discomfort which has a direct impact on the compliance and quality of life of patients. Many pharmacological methods over the past years have been recommended to ease the pain and discomfort and make orthodontic treatment more acceptable .These methods have adverse effects and hence it would be beneficial if we propose a method which will satisfy the patients and will be suitable for them to follow with minimal side effects and maximum efficacy.

Null hypothesis: lignocaine gel and chewing gum will be equally effective in reducing pain after separator placement Alternative hypothesis: lignocaine gel will be more effective than chewing gum in reducing pain after separator placement

DETAILED DESCRIPTION:
Data will be collected from subjects reporting to the department of orthodontics, Karachi Medical and Dental College. This study will be started after submission of the synopsis and after approval of the Ethical Review Committee.

Following the placement of separators participant will be randomly assigned in to 2 groups.It is a parallel group randamization.In this study the topical gel (lignocaine ) and a sugar free gum that is commercially available is purchased from the local market. The composition of lignocaine gel is given .Manual allocation using sealed envelope during enrolment of patient in the study. This enabled approximately equal distribution of patients from each group.

1. st group: Topical gel (lignocaine gel)
2. nd group: chewing gum In our study all the participant were asked to fill the questionnaire. A written informed consent was acquired from all patients for inclusion in the study.

In the topical gel group the patients were directed to apply the gel on the buccal free gingival margin of their first molar at one side when the separators are placed and reapply the gel every 8 hours . They were then requested to mark their level of pain at 2 and 8 hours and at 10 pm of the 2nd,3rd,5th and 7th day after the gel is being applied and mark it on the VAS form.

The patients in the chewing gum group were advised to chew sugar free gum for 5 minutes immediately after separators were placed and at 8 hours interval. The patients were also advised and motivated not to take any additional analgesics.

For measuring the perception of pain the most reliable method is the Visual Analog Scale (VAS).It is a psychometric pain response scale.VAS is a measurement instrument for subjective characters such as pain which cannot be measured directly.

The VAS form was filled in by the patients at baseline after separator placement at 2 hours, at 8 hours , 24 hours, at 2nd day , 3rd day , 5th and 7th day after separator placement. When replying to the VAS performa , the patients were requested to state their severity of pain by marking a position along a calibrated straight continous line weighted at both ends by descriptive terminology with a happy face and a sad face and document the severity of pain when the jaws are at rest and during the biting activity.The degree of pain was determined solely , based on patients conviction through VAS cards and questionnaire .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy with no significant medical finding
2. Currently not taking antibiotics or analgesics
3. No contraindication to the use of chewing gum/topical analgesics
4. Minimum age 12 years ,maximum age 30 years
5. Literate/English speaking

Exclusion Criteria:

1. Patient who did not return the completed questionnairs
2. Using analgesics or antibiotics

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-03-12 (Estimated); Study Completion 2023-03-16 (Estimated)

PRIMARY OUTCOMES:
pain reduction | 2 hours, at 8 hours , 24 hours, at 2nd day , 3rd day , 5th and 7th day after separator placement.
  Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Sadaf Bashir, BDS, Principal Investigator — Karachi Medical and Dental College
Locations (1):
- Sadaf Bashir, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
response to each variable of the questionnaire, name, age , occupation,gender,
Supporting Information: Study Protocol, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: Sadaf bashir